CLINICAL TRIAL: NCT01369745
Title: A Phase II, Double-Blind, Placebo-Controlled, Multi-Center, Randomized Withdrawal Design Trial Using Adaptive Randomization Comparing Z-102 With Placebo In Patients With Moderate To Severe Rheumatoid Arthritis
Brief Title: A Phase II Trial Comparing Z-102 With Placebo In Patients With Moderate To Severe Rheumatoid Arthritis
Acronym: Synergy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zalicus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Z102-008
Record Dates: First submitted 2011-06-07; First posted 2011-06-09 (Estimated); Results first posted 2014-04-30 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Moderate to severe
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Prednisolone; Dipyridamole; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Prednisolone (Active Comparator): Prednisolone 2.7 mg daily for 12 weeks
  Interventions: Drug: Prednisolone
- dipyridamole (Active Comparator): Dipyridamole 360 mg daily for 12 weeks
  Interventions: Drug: dipyridamole
- prednisone (Active Comparator): Prednisone 5 mg daily for 12 weeks
  Interventions: Drug: Prednisone
- Z102 (2.7/360) (Experimental): Prednisolone 2.7 mg plus dipyridamole 360 mg daily for 12 weeks
  Interventions: Drug: Z102
- placebo (Placebo Comparator): Placebo daily for 12 weeks
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Prednisolone — Prednisolone 2.7 mg daily
  Arms: Prednisolone
Drug: dipyridamole — dipyridamole 360 mg daily
  Arms: dipyridamole
Drug: Prednisone — Prednisone 5 mg daily
  Arms: prednisone
Drug: Z102 — Prednisolone 2.7 mg plus dipyridamole 360 mg daily
  Other Names: prednisolone; dipyridamole
  Arms: Z102 (2.7/360)
Other: placebo
  Arms: placebo

SUMMARY:
Thus study will test an experimental drug called Z-102 (combination of prednisolone and dipyridamole) to treat patients with moderate to severe rheumatoid arthritis.

DETAILED DESCRIPTION:
The primary objective of the study was to demonstrate the efficacy of Z102 (2.7 mg prednisolone/360 mg dipyridamole) versus placebo on the Disease Activity Score 28 using C reactive protein (DAS28-CRP) in subjects with rheumatoid arthritis at the study endpoint of 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Meet the ACR / EULAR criteria for classification of RA
* Have moderate to severe RA, defined as involving a minimum (≥6 total swollen and ≥6 total tender) of the 28 joints assessed
* Have screening CRP levels of at least 0.6 mg/dl and a DAS28-CRP score ≥4.5
* Have been on a stable dose of conventional DMARD therapy for at least 90 days without dosage adjustment or modification and should be able to maintain the same dose of conventional DMARD therapy during study participation (with or without glucocorticoid therapy

Exclusion Criteria:

* Treatment-refractory patients are excluded
* Has active cardiovascular disease, unless well controlled by appropriate treatment for a minimum of 3 months prior to screening
* Is taking aspirin for reasons other than for cardiovascular prophylaxis or their total daily dose is greater than 325 mg
* Is currently taking steroids at a daily prednisone dose, or the equivalent, of >10 mg
* Intraarticular, intramuscular, or intravenous glucocorticoids must not have been given at least 6 weeks prior to entering the study
* The need to continue the use of one or multiple NSAID's at the same time, or the use of acetaminophen on a chronic basis
* All opiate use is prohibited
* Use of any other medications or herbs used for the treatment of pain is prohibited
* Patients with a history of or currently active tuberculosis as per specific country guidelines are excluded
* Has uncontrolled diabetes mellitus as defined by a serum glucose >126 mg/dl
* Knowingly has HIV infection or hepatitis
* Has undergone administration of any investigational drug within 30 days of study initiation
* All biologic agents are excluded for 90 days prior to Screening and throughout the study.
* Has undergone administration of rituximab or any B-cell depleting investigational drugs within 6 months of study initiation
* Has had a history of alcohol or drug abuse within the past 2 years
* Has a history of hypersensitivity to glucocorticoids and/or dipyridamole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Lee, PhD, Study Director — Zalicus, Inc.
Locations (1):
- Zalicus Investigational Site, Toledo, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 294 subjects entered the titration phase. Of these, 258 subjects completed the titration phase, were randomized to treatment, received at least one dose of study drug and constitute the safety population. Of these, 252 subjects provided at least one post-baseline measurement of the primary endpoint and constitute the efficacy population.
Groups:
- Prednisolone: Prednisolone 2.7 mg once daily
- Dipyridamole: dipyridamole 360 mg once daily
- Prednisone: Prednisone 5 mg once daily
- Z102: 2.7 mg prednisolone plus 360 mg dipyridamole once daily
- Placebo: placebo once daily
Period: Overall Study
Arm/Group | Prednisolone | Dipyridamole | Prednisone | Z102 | Placebo
Started | 32 | 41 | 18 | 84 | 83
Completed | 25 | 28 | 16 | 64 | 65
Not Completed | 7 | 13 | 2 | 20 | 18

BASELINE CHARACTERISTICS:
Population: population randomized to double blind phase of study and recieved at least one dose of study drug
Groups:
- Prednisolone: Prednisolone 2.7 mg once daily The trial would progress from Stage 1 to Stage 2 if the posterior probability that Z102 is superior to placebo was greater than 0.975.
- Dipyridamole: dipyridamole 360 mg once daily The trial would progress from Stage 2 to Stage 3 if the posterior probability that Z102 is superior to dipyridamole was greater than 0.975.
- Prednisone: Prednisone 5 mg once daily The trial would progress from Stage 2 to Stage 4 if the posterior probability that Z102 is superior to prednisolone 2.7 was greater than 0.975.
- Z102: prednisolone 2.7 mg plus dipyridamole 360 mg once daily The trial would progress from Stage 3 to Stage 5 if the posterior probability that Z102 is superior to prednisolone 2.7 was greater than 0.975.
- Total: Total of all reporting groups
Arm/Group | Prednisolone | Dipyridamole | Prednisone | Z102 | Placebo | Total
Number analyzed (Participants) | 32 | 41 | 18 | 84 | 83 | 258
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (12.69) | 55.9 (9.35) | 55.5 (9.82) | 54.5 (11.53) | 53.7 (12.44) | 54.6 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 36 | 17 | 72 | 75 | 226
  Male | 6 | 5 | 1 | 12 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in DAS28-CRP at 12 Weeks
Description: The primary efficacy endpoint was the mean change in Disease Activity Score 28 using C-reactive protein (DAS28-CRP) from baseline to Week 12.
  The DAS28-CRP is a composite measure of inflammation in Rheumatoid Arthritis and incorporates a tender and swollen joint count, CRP and Patient Global Assessment of Disease Activity expressed in a Gaussian distribution of variables ranging from 0 to 10. A DAS28-CRP score of <3.2 suggests a low level of disease activity, while a score of >5.1 suggests a high level of disease activity. Using the DAS-CRP as a continuous scale allows investigators (and clinicians) to measure a clinically meaningful endpoint following institution of a therapeutic intervention. In RA, clinical remission would therefore be graded as a DAS28 score of ≤3.2 with disease flare accompanying scores of ≥5.1; well-controlled disease is best characterized as fitting in between these two scores.
Time Frame: baseline to week 12
Population: The efficacy analysis population includes all 252 subjects who received at least one dose of study drug after randomization and who provided at least one post-baseline measurement of the primary endpoint
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Z102: prednisolone 2.7 mg plus dipyridamole 360 mg once daily
Arm/Group | Prednisolone | Dipyridamole | Prednisone | Z102 | Placebo
Number analyzed (Participants) | 32 | 39 | 18 | 82 | 81
units on a scale | -1.147 (0.235) | -0.813 (0.216) | -1.237 (0.296) | -0.907 (0.149) | -0.538 (0.153)

2. Secondary Outcome: Change From Baseline in DAS28-CRP Individual Components at 12 Weeks
Description: The mean change in the individual components of the Disease Activity Score 28 using C-reactive protein (DAS28-CRP) from baseline to Week 12 which included individual assessment of Tender Joint Count (28-joint assessment), Swollen Joint Count (28-joint assessment), Patient Global Assessment of Disease Activity and absolute CRP level. In each case, higher scores indicate more disease activity.
  The DAS28-CRP is a composite measure of inflammation in Rheumatoid Arthritis and incorporates a tender and swollen joint count, CRP and Patient Global Assessment of Disease Activity expressed in a Gaussian distribution of variables ranging from 0 to 10. A DAS28-CRP score of <3.2 suggests a low level of disease activity, while a score of >5.1 suggests a high level of disease activity.
Time Frame: Baseline to week 12
Population: Because the study never progressed past the first stage of the adaptive randomization, the number of subjects who were allocated to the dipyridamole 360 mg, prednisolone 2.7 mg, and prednisone 5 mg treatment arms was insufficient (underpowered) to allow analysis of the secondary objectives.
Arm/Group | Prednisolone | Dipyridamole | Prednisone | Z102 | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Percentage of Subjects Achieving ACR20, ACR50 and ACR70 at 12 Weeks
Description: The American College of Rheumatology (ACR) 20 is a widely accepted composite index of improvement in RA proposed by the ACR (Fransen and van Riel 2009). ACR20 refers to a composite improvement of 20% in swollen joint count, tender joint count, and 3 or more of the following 5 measures:Physician's Global Assessment of Disease Activity, Patient's Global Assessment of Disease Activity, Patient Pain VAS, Patient's self-addressed disability (HAQ) (Arnet 1988 and Felson 1995), Acute-phase reactant (ESR or CRP) The ACR 50 and ACR 70 are similar tools, used to indicate 50% and 70% improvement, respectively.
Time Frame: Week 12
Population: as for outcome 2
Arm/Group | Prednisolone | Dipyridamole | Prednisone | Z102 | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Multidimensional Assessment of Fatigue (MAF) at Week 12
Description: The Multidimensional Assessment of Fatigue (MAF) scale contains 16 items and measures four dimensions of fatigue: severity (#1-2), distress (#3), degree of interference in activities of daily living (#4-14), and timing (#15-16). Fourteen items contain numerical rating scales (#1-14) and two items have multiple-choice responses (#15-16). Respondents are asked to reflect on fatigue patterns for the past week.
  To calculate the Global Fatigue Index (GFI): Convert item #15 to a 0-10 scale by multiplying each score by 2.5 and then sum items #1, 2, 3, average #4-14, and newly scored item #15.
  Scores range from 1 (no fatigue) to 50 (severe fatigue). Do not assign a score to items #4-14 if respondent indicated they "do not do any activity for reasons other than fatigue." If respondents select no fatigue on item #1, assign a zero to items #2-16. Item #16 is not included in the Global Fatigue Index.
Time Frame: week 12
Population: as for outcome 2
Arm/Group | Prednisolone | Dipyridamole | Prednisone | Z102 | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Time to Failure (Days)
Description: Patients will be monitored for addition of any DMARD or withdrawal due to flare. The time to failure is defined as the duration of study participation (in days) until a qualifying event or completion of study treatment, whichever comes first.
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Arm/Group | Prednisolone | Dipyridamole | Prednisone | Z102 | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of consent through the end of study visit at 12 weeks.
Description: Adverse events are reported for the safety population of 258 subjects randomized to the double blind study phase and who received at least one dose of study drug.
Arm/Group | Prednisolone | Dipyridamole | Prednisone | Z102 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/32 | 2/41 | 0/18 | 5/84 | 4/83
Other Adverse Events (participants affected / at risk) | 6/32 | 30/41 | 5/18 | 38/84 | 33/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prednisolone (N=32) | Dipyridamole (N=41) | Prednisone (N=18) | Z102 (N=84) | Placebo (N=83)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureteric Obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus Ureteric (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prednisolone (N=32) | Dipyridamole (N=41) | Prednisone (N=18) | Z102 (N=84) | Placebo (N=83)
Headache (Nervous system disorders) | 1 | 11 | 0 | 13 | 4
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 5 | 8
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 5 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 1 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 1
Abdominal Upper Pain (Gastrointestinal disorders) | 1 | 3 | 0 | 1 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1 | 1 | 4
Rash Pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 2
Oedema Peripheral (General disorders) | 1 | 0 | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
The study did not progress past the first stage of adaptive randomization. The number of subjects allocated to the dipyridamole 360 mg, prednisolone 2.7 mg, and prednisone 5 mg arms was insufficient to allow analysis of the secondary objectives.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less